CLINICAL TRIAL: NCT04853147
Title: Triple Combination of Fosaprepitant, Dexamethasone and Palonosetron Versus Combination of Dexamethasone and Palonosetron for the Prevention of Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Gastrointestinal Surgery
Brief Title: Triple Therapy for Postoperative Nausea and Vomiting in Laparoscopic Gastrointestinal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, YangZhao, deputy director, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: E2020170
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: C.Surgical Procedure; Gastrointestinal
Keywords: postoperative nausea and vomiting, fosaprepitant,
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Palonosetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- triple therapy (Experimental): Triple combination of Fosaprepitant, Palonosetron and Dexamethasone were administered
  Interventions: Drug: palonosetron, dexamethasone, and fosaprepitant dissolved in 0.9% NaCl
- double therapy (Other): double combination of Palonosetron and Dexamethasone were administered
  Interventions: Drug: palonosetron, dexamethasone, and 0.9% NaCl

INTERVENTIONS:
Drug: palonosetron, dexamethasone, and fosaprepitant dissolved in 0.9% NaCl — palonosetron 0.075 mg, iv, dexamethasone 5mg, iv, fosaprepitant 150mg dissolved in 0.9% NaCl 150ml, iv.drip,
  Other Names: Triple therapy
  Arms: triple therapy
Drug: palonosetron, dexamethasone, and 0.9% NaCl — palonosetron 0.075 mg, iv, dexamethasone 5mg, iv, 0.9% NaCl 150ml, iv.drip,
  Other Names: double therapy
  Arms: double therapy

SUMMARY:
Postoperative nausea and vomiting (PONV) are common in patients, especially in patients at high risk. PONV may result in prolonged hospital stay and threaten patients' life. Because the etiology of PONV is very complex, there is an increasing focus on combining antiemetics from different classes for PONV prophylaxis. Fosaprepitant is a neurokinin-1 (NK-1) receptor antagonist to prevent PONV. Palonosetron is a 5-HT3 receptor antagonist with high efficacy and sustained action for PONV prophylaxis. Dexamethasone belongs to corticosteroid and also has the ability to reduce the incident of PONV. This study aims to use the combination of these three drugs in high-risk patients to test whether triple therapy is better than combination of palonosetron and dexamethasone to prevent PONV.

DETAILED DESCRIPTION:
This trial is a prospective, randomized controlled study with blinded participant, care provider, investigator, and outcomes assessor. 1154 patients aged 18 to 75 years undergoing laparoscopic gastrointestinal surgery will be enrolled.Triple therapy of palonosetron and dexamethasone plus fosaprepitant will be administered in the intervention group, and double therapy of palonosetron and dexamethasone will be used in the control group. The anxiety of patients will be evaluated. The primary outcome is proportion of participants with PONV during the first 24 postoperative hours. Secondary outcomes are as follow: proportion of participants with PONV,emetic episodes, nausea, with rescue antiemetic medication; the scores of QOR-15; pain scores;time to first flatus after surgery; time to first defecation after surgery; recovery time; health related quality of life; proportion of participants with adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and Age ≤75 years;
* Scheduled for laparoscopic gastrointestinal surgical procedure with general anesthesia ;
* The score evaluated by Apfel simplified PONV risk assessment systems is ≥3.

Exclusion Criteria:

* The American Society of Anesthesiologists (ASA) rating is >3;
* Severe hepatic dysfunction(the score of Child-Pugh is >9);
* With contraindications for using fosaprepitant, 5-HT3 receptor antagonist or dexamethasone ;
* Take medications with known antiemetic properties preoperatively ;
* With mental disorder, or not be able to communicate ;
* Pregnant women or nursing mothers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1154 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with PONV during the first 24 postoperative hours | from operation completion to 24-hour after surgery (up to 24 hours)
  PONV is defined as nausea, retching or vomiting

SECONDARY OUTCOMES:
Proportion of participants with PONV | calculated at 24-hour, 72-hour, 120-hour after surgery(daily recorded up to 120 hours after surgery)
  PONV is defined as nausea, retching or vomiting
Proportion of participants with emetic episodes | calculated at 24-hour, 72-hour, 120-hour after surgery(daily recorded up to 120 hours after surgery)
  Emetic episodes are defined as retching or vomiting or both
Proportion of participants with nausea | calculated at 24-hour, 72-hour, 120-hour after surgery(daily recorded up to 120 hours after surgery)
  Nausea is defined as a feeling of the urge to vomit
Proportion of participants with rescue antiemetic medication | calculated at 24-hour, 72-hour, 120-hour after surgery(daily recorded up to 120 hours after surgery)
  Rescue antiemetic medication
The severity of PONV | calculated at 24-hour, 72-hour, 120-hour after surgery(daily recorded up to 120 hours after surgery)
  The severity of PONV is evaluated by a PONV impact scale score. Nausea intensity is scored as 1 ,2 ,3. In addition, vomiting intensity is scored as the number of vomits (0-2, or 3 if three or more vomits). Both scores together to obtain the PONV impact scale score
Postoperative recovery score using 15-item quality of recovery scoring system(QoR-15) during each subsequent evaluation period (up to 120 hours) | evaluated at 24-hour, 72-hour, 120-hour after surgery(up to 120 hours after surgery)
  The QoR-15 comprises five subscales: pain, physical comfort, physical independence, psychological support, and emotional state. Each item is scored from 0 to 10, and the possible total score ranges from 0 to 150. A higher total score means better patient QoR.
Pain scores | evaluated at 24-hour, 72-hour, 120-hour after surgery(up to 120 hours after surgery)
  Pain scores are evaluated by numerical rating scale(NRS) from no pain(0) to most severe pain (10).
Time to first flatus after surgery | evaluated at the time of first exhaust after surgery(expected average of 3 days after surgery)
  Time length between operation completion and the first flatus
Time to first defecation after surgery | evaluated at the time of the first defecation after surgery(expected average of 6 days after surgery
  Time length between operation completion and the first defecation
Time to fulfill the criteria of hospital discharge (recovery time) | from operation completion to fulfill the criteria of hospital discharge(expected 6 days )
  The ideal time point for discharge, which is also considered as recovery time.
Health related quality of life | evaluated before surgery, at 120-hour and 30 days after surgery (up to 30 days）
  Health related quality of life is measured by EQ-5D. Each EQ-5D health state can be coded into a five-digit number using the numbers 1 , 2 , and 3 to indicate the functional levels of the five dimensions.
Proportion of patients with adverse events (up to 30 days after surgery) | from drug administration to 30 days (30 days)
  adverse events

OTHER OUTCOMES:
Concentration of materials in blood such as hormone and metabolic | evaluated before surgery, at the end of surgery
  materials in blood
6-month survival rate | 6-month after surgery
  survival rate in 6-month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yang Zhao, Doctor, Principal Investigator — Sixth SunYetSen
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moon HY, Baek CW, Choi GJ, Shin HY, Kang H, Jung YH, Woo YC, Kim JY, Park SG. Palonosetron and aprepitant for the prevention of postoperative nausea and vomiting in patients indicated for laparoscopic gynaecologic surgery: a double-blind randomised trial. BMC Anesthesiol. 2014 Aug 10;14:68. doi: 10.1186/1471-2253-14-68. eCollection 2014. PMID 25165427
- [Background] Lim CS, Ko YK, Kim YH, Park SI, Kim JK, Kim MJ, Kim HJ. Efficacy of the oral neurokinin-1 receptor antagonist aprepitant administered with ondansetron for the prevention of postoperative nausea and vomiting. Korean J Anesthesiol. 2013 Mar;64(3):212-7. doi: 10.4097/kjae.2013.64.3.212. Epub 2013 Mar 19. PMID 23560185
- [Background] DREAMS Trial Collaborators and West Midlands Research Collaborative. Dexamethasone versus standard treatment for postoperative nausea and vomiting in gastrointestinal surgery: randomised controlled trial (DREAMS Trial). BMJ. 2017 Apr 18;357:j1455. doi: 10.1136/bmj.j1455. PMID 28420629
- [Background] Rojas C, Stathis M, Thomas AG, Massuda EB, Alt J, Zhang J, Rubenstein E, Sebastiani S, Cantoreggi S, Snyder SH, Slusher B. Palonosetron exhibits unique molecular interactions with the 5-HT3 receptor. Anesth Analg. 2008 Aug;107(2):469-78. doi: 10.1213/ane.0b013e318172fa74. PMID 18633025
- [Background] Gouveia de Araujo Ferreira N, Cavalcanti IL, Assad AR, Barrucand L, Braga ELC, Vercosa N. A prospective, randomized, double-blind trial to compare body weight-adjusted and fixed doses of palonosetron for preventing postoperative nausea and vomiting in obese female patients. PLoS One. 2020 Jan 14;15(1):e0227490. doi: 10.1371/journal.pone.0227490. eCollection 2020. PMID 31935249
- [Background] Wang EHZ, Sunderland S, Edwards NY, Chima NS, Yarnold CH, Schwarz SKW, Coley MA. A Single Prophylactic Dose of Ondansetron Given at Cessation of Postoperative Propofol Sedation Decreases Postoperative Nausea and Vomiting in Cardiac Surgery Patients: A Randomized Controlled Trial. Anesth Analg. 2020 Oct;131(4):1164-1172. doi: 10.1213/ANE.0000000000004730. PMID 32925337
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Amirshahi M, Behnamfar N, Badakhsh M, Rafiemanesh H, Keikhaie KR, Sheyback M, Sari M. Prevalence of postoperative nausea and vomiting: A systematic review and meta-analysis. Saudi J Anaesth. 2020 Jan-Mar;14(1):48-56. doi: 10.4103/sja.SJA_401_19. Epub 2020 Jan 6. PMID 31998020
- [Background] Hooper VD. SAMBA Consensus Guidelines for the Management of Postoperative Nausea and Vomiting: An Executive Summary for Perianesthesia Nurses. J Perianesth Nurs. 2015 Oct;30(5):377-82. doi: 10.1016/j.jopan.2015.08.009. No abstract available. PMID 26408511
- [Background] Apfel CC, Heidrich FM, Jukar-Rao S, Jalota L, Hornuss C, Whelan RP, Zhang K, Cakmakkaya OS. Evidence-based analysis of risk factors for postoperative nausea and vomiting. Br J Anaesth. 2012 Nov;109(5):742-53. doi: 10.1093/bja/aes276. Epub 2012 Oct 3. PMID 23035051
- [Derived] Huang Q, Wang F, Liang C, Huang Y, Zhao Y, Liu C, Lin C, Zhang L, Zhou S, Wang Q, Li S, Gong R, Wu Q, Gu Y, Zhang J, Luo T, Wang W, Zhang S, Bizo Mailoga N, Wang K, Jin S, Zhao Y. Fosaprepitant for postoperative nausea and vomiting in patients undergoing laparoscopic gastrointestinal surgery: a randomised trial. Br J Anaesth. 2023 Oct;131(4):673-681. doi: 10.1016/j.bja.2023.06.029. Epub 2023 Jul 7. PMID 37423834

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT04853147/Prot_SAP_000.pdf